CLINICAL TRIAL: NCT05745051
Title: A Single-center, Clinical Trial to Evaluate the Safety and Effectiveness of CVA-FLOW Software Device for Acute Ischemic Stroke
Brief Title: The Safety and Effectiveness of CVA-FLOW Software Device for Acute Ischemic Stroke
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cvaid Medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 0091-22-SZMC
Record Dates: First submitted 2023-02-07; First posted 2023-02-27 (Actual); Last update posted 2023-08-30 (Actual); Status verified 2023-08

CONDITIONS: Stroke; Stroke, Acute; Stroke, Ischemic; Stroke, Cardiovascular; Stroke Hemorrhagic
MeSH Terms: conditions — Stroke; Ischemic Stroke; Myocardial Infarction; Hemorrhagic Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Evaluate the safety and effectiveness of CVA-FLOW Software Device for acute ischemic stroke (Experimental): The purpose of this study is to demonstrate the effectiveness and safety of CVA-FLOW, a digital health AI based Telestroke system developed by CVAID Ltd. Company aims to assist certified medical staff to triage acute ischemic stroke patients using dedicated algorithms in order to support application for market approval for CVA-FLOW device.
  Interventions: Diagnostic Test: CVAid Flow

INTERVENTIONS:
Diagnostic Test: CVAid Flow — CVA-FLOW is a Telestroke mobile software solution that enables the neurologist to remotely assess, on his smartphone, patients suspected with stroke. Real-time, objective, patient-specific data such as images, videos and vocal records of the patient, are acquired by a first responder (CVA-COLLECTOR) at the patient's location. This allows the neurologist to complete the NIH Stroke Scale and independently reach a diagnostic conclusion and treatment plan (CVA-MED).

SUMMARY:
The purpose of this study is to demonstrate the effectiveness and safety of CVA-FLOW, a digital health AI based Telestroke system developed by CVAID Ltd. Company aims to assist certified medical staff to triage acute ischemic stroke patients using dedicated algorithms in order to support application for market approval for CVA-FLOW device.

ELIGIBILITY:
Inclusion Criteria:

* Suspected hyper-acute stroke patient at the ED, prior to treatment (tPA or EVT)
* Age≥18

Exclusion Criteria:

* Intubated patients upon arrival
* Time from stroke symptoms onset > 24h
* Patients post treatment (tPA of EVT)
* Patient in acute psychosis state
* Patients who do not speak Hebrew as their mother tongue

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-11-08 (Actual); Primary Completion 2023-10-30 (Estimated); Study Completion 2023-11-30 (Estimated)

PRIMARY OUTCOMES:
Sensitivity and specificity of stroke severity classification by CVA-CORE algorithm | At admission
  Stroke severity classification will be calculated by the CVA-CORE system algorithm and compared to the imaging results (interpretation).
Sensitivity and specificity of stroke severity classification by CVA-CORE algorithm | after 24 hours
  Stroke severity classification will be calculated by the CVA-CORE system algorithm and compared to the imaging results (interpretation).

SECONDARY OUTCOMES:
Device operational performance | At admission
  The investigator shall assess the use of the device during the operation, and conclude a summary evaluation after the end of the usage. Evaluation items are shown below:Item / evaluation
  * Usage experience: Simple to operate/difficult to operate
  * Errors: No errors occurs during the usage/ Errors occurs during the usage
  * Known safety issues during use of CVA-MED and CVA-COLLECTOR
Device operational performance | after 24 hours
  The investigator shall assess the use of the device during the operation, and conclude a summary evaluation after the end of the usage. Evaluation items are shown below:Item / evaluation
  * Usage experience: Simple to operate/difficult to operate
  * Errors: No errors occurs during the usage/ Errors occurs during the usage
  * Known safety issues during use of CVA-MED and CVA-COLLECTOR

CONTACTS AND LOCATIONS:
Locations (1):
- Shaare Zedek Medical Center, Jerusalem, Israel

IPD SHARING:
Plan to Share IPD: No